CLINICAL TRIAL: NCT06550414
Title: Effect Of Use of Dexmedetomidine as an Adjuvant to Bupivacaine 0.1% in Labor Analgesia.
Brief Title: Dexmedetomidine As An Adjuvant To Bupivacaine 0.1% in Labor Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Services Institute of Medical Sciences, Pakistan (Other Government)
Responsible Party: Principal Investigator, dr. sana siddiq, assistant professor, Services Institute of Medical Sciences, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HLH
Record Dates: First submitted 2024-08-05; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Labor Analgesia; Labor Pain
Keywords: bupivacaine; Dexmedetomidine; Labor analgesia
MeSH Terms: conditions — Labor Pain | interventions — Dexmedetomidine; Bupivacaine

STUDY DESIGN:
Intervention Model Description: randomized control trial
Who Masked: Investigator
Masking Description: double blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- bupivacaine group (Placebo Comparator): group given 0.1% bupivacaine 10ml as loading dose in labor epidural.
  Interventions: Drug: Bupivacain
- dexmedetomidine group (Active Comparator): group given 50 micrograms of dexmedetomidine along with 0.1% bupivacaine in labor analgesia dose.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Active comparator: dexmedetomidine group
  Other Names: Labor analgesia
  Arms: dexmedetomidine group
Drug: Bupivacain — Placebo comparator: bupivacaine group
  Other Names: Labor analgesia
  Arms: bupivacaine group

SUMMARY:
Females who have experienced normal labor for child birth have claimed it to be most difficult and distressing moments of their life due to excruciating and unbearable pain. Provision of effective and satisfactory labor analgesia to the parturient helps in achieving greater degree of well-being for both mother and child. Several medical and non-medical pain relief methods are used since ages for pain relief during childbirth.

Epidural anesthesia and intravenous opioids (pethidine) are most commonly offered to the mothers for relieving labor pain. So far, Epidural is considered gold standard in attaining maternal satisfaction for pain free deliveries. lt can be modified for individual parturient in order to achieve highest level of comfort and pain relief. To attain better and prolonged analgesia several additives have been used with local anesthetists and their effects are studied. Epidural opioids are conventionally being used as adjuvants, however associated side effects (nausea, vomiting, and pruritus) may limit their use. An alpha 2 adrenoceptor agonist, dexmedetomidine, has been effectively used and studied in labor epidurals and provided better analgesia without significant side effects. Hamed Lateef Hospital is one of the largest tertiary care private setup offering painless deliveries in Lahore.

It is need of the hour to modify and improve our clinical practice in order to achieve highest level of patient satisfaction and provision of best possible maternal and fetal outcome. This study is proposed to investigate and elaborate the effect of adding dexmedetomidine to bupivacaine in labor epidurals and to study possible side-effects associated with its use.

DETAILED DESCRIPTION:
Objectives of this study are to evaluate the efficacy of adding dexmedetomidine in labor epidurals with 0.1% bupivacaine in females undergoing normal vaginal delivery.

OPERATIONAT DEFINITIONS:

1. Onset of Analgesia:

   Time required to attain a VAS of less than or equal to 3 after giving loading dose
2. Duration of Analgesia. Time after loading dose till the VAS >3 or break-through pain reported by the mother.
3. Side effects:

   * Hypotension: systolic blood pressure < 100 mmHg or a decrease in mean arterial pressure (MAP) > 30% compared to the baseline
   * Bradycardia: heart rate less than 60.
   * Nausea, vomiting
   * Sedation

HYPOTHESIS:

Duration of Analgesia is prolonged and onset of analgesia is shortened after adding dexmedetomidine with bupivacaine without any significant side effects.

STUDY DESIGN:

Prospective double blinded randomized control trial.

SETTING:

This prospective randomized control trial will be conducted at the Department of anesthesiology Hamed Latif Hospital in six months after approval from local ethical committee.

SAMPLE SIZE:

Sample size is calculated using G power software. Keeping Alpha error 0.05 and power of study 80% the total sample size is calculated to be 134 It is equally divided in 2 groups. This study is proposed for the pregnant females in active labor in obstetrical and gynecological department of Hamed Latin Hospital who request epidural analgesia for pain relief during normal vaginal delivery.

SAMPLING TECHNIQUE:

Non probability purposive sampling.

Sample selection:

INFORMED CONSENT:

Before participating in the study, all cases will be informed about the benefits and risks of epidural analgesia along with the medications used. A written informed consent will be obtained after that.

MATERIALS AND METHODS:

DATA COILECTION PROCEDURE:

The closed envelope opened after randomization with the computer-generated method will be used to randomly divide the patient in each group.

The included 134 women will be equally allocated into two groups:

Control group (64 women) which will receive bupivacaine 0.1% (10 ml) in normal saline, and dexmedetomidine group (64 women) that will receive the same amount of bupivacaine in addition to dexmedetomidine 50 microm in normal saline as a loading dose (5 ml increments/s min). This will be followed by continuous infusion of bupivacaine 0.1% (at 10 ml/h rate) for both groups, which will be stopped with full cervical dilatation. The epidural solutions will be prepared by an anesthesiologist not included in the study. Moreover, all of the following will be blinded: A) Anesthesiologist giving epidural analgesia. B) Resident following labor progress and pain scoring. All of the included women (in an active second stage of labor with cervical dilatation of 3-5 cm) will be give Hartman's solution (500 ml) as a preload; then, routine baseline monitoring will be started including blood pressure (non-invasive), electrocardiography, and pulse oximetry. Also, they will be explained how to report their pain degree according to the visual analog scale (VAS) (0 for no pain felt at all, to 10 for the worst pain ever felt). After that they will be placed in the sitting position with proper sterilization of the back, followed by local infiltration of the skin with underlying subcutaneous tissue overlying lumbar (L) 3-4 and L 4-5 intervertebral disc by lidocaine 2%.The epidural space will be reached via an 18- gauge needle, and this will be ensured using the loss of resistance to air technique. Next, aspiration will be done to exclude the presence of blood or cerebrospinal fluid followed by injection of 3 ml of lidocaine 2% as a test dose. After that, a 2O-gauge multi-orifice epidural catheter will be introduced and fixed at 4.5-5.5 depth. Catheter will be secured and woman will be placed in lateral position to avoid compression of the inferior cavil vein by the pregnant uterus. Injection of the study solution will be given only in between uterine contractions to decrease the risk of drug overspread in the epidural space. lf VAS>3 or break-through pain will be reported by the patient then a top-up dose of bupivacaine 0.1% (10 ml)will be given' The top up doses number will be recorded. The modified Bromage scale will be used to assess the degree of motor block before installation of the epidural catheter, every 15 min during the 1st hour after installation and then every 30 min till delivery.

lf Bromage score > 2 will be detected, bupivacaine infusion rate will be decreased till achieving a score less than 3.

1. Side effects will be reported and managed according. Both heart rate and arterial blood pressure will be monitored and recorded before the installation of the epidural catheter, and 5, 15, 30,45, and 60 min following its installation and then hourly till the end of delivery. Hypotension, defined as systolic blood pressure < 100 mmHg or a decrease in mean arterial pressure (MAP) > 30% compared to the baseline, and will be managed by Phenylephrine (bolus of 50 micrograms) along with intravenous fluids. Bradycardia, defined as heart rate (HR) less than 60 beats/m, and will be managed by intravenous 0.5 mg atropine' Cardiotocography will be used for fetal heart rate monitoring. lf any abnormalities will be detected, the mother will be asked to change her position to the left lateral one. The time needed for cervical dilatation, the duration of each stage of labor, and the mode of delivery will recorded. After 6 h of delivery, mother satisfaction will be assessed with the five-point Likert's scale as follows: 1 for poor, 2 for fair,3 for good, 4 for very good, and 5 for excellent satisfaction. The primary outcome will be the onset of analgesia, while the secondary outcomes include the duration of analgesia, hemodynamic changes, labor progress, and maternal complications. Data will be entered, tabulated and analyzed using SPSS, version 26. After data entering baseline characteristics will be described as frequencies and percentages, mean values and standard deviation (SD), or median and range. For comparison of two independent groups of qualitative data, Chi-Square test (or Fisher's exact test) will be applied. Besides, Mann-Whitney U test and independent-samples test will be used to compare two groups of non-parametric and parametric quantitative data respectively. P values < 0.05 will be considered statistically significant for all of the used statistical tests

ELIGIBILITY:
Inclusion Criteria:

* Patients in 37 or more weeks of pregnancy,
* having a single pregnancy with vertex presentation
* without any significant systemic disease will be included in the study.

Exclusion Criteria:

* Patients with mal-presentation
* twin pregnancy
* preeclampsia,
* uncontrolled systemic comorbidities
* diabetes, renal, hepatic, or cardiac.
* bleeding, diathesis, body mass index (BMl) more than 35 kg/m2
* known allergy to any of the study drugs will be excluded from the study.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 37 weeks or more pregnant female in active labor.
Enrollment: 165 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
onset of analgesia | Patient observed for 45 minutes after drug delivery and time required to achieve a VAS of 3 or less than 3 is noted down.
  time noted for onset of analgesia in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Siddiq, Principal Investigator — Hameed lateef hospital
Locations (1):
- Hameed Lateef Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No